CLINICAL TRIAL: NCT04284306
Title: Immunohistochemical Assessment of Programmed Death Ligand 1 PDL-1 and Autophagy Marker LC3B in Glioblastoma
Brief Title: Immunohistochemical Assessment of Programmed Death ligand1 and LC3B in GBM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana Fathy Ali Torky, Assissant lecturer,Department of Pathology,Faculty of medicine Assiut university, Assiut University
Other Study IDs: PDL-1 and LC3B in GBM
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Glioblastoma Multiforme
Keywords: PDL-1; LC3B
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Formaline-fixed-paraffin-embedded tissue specimens .
Oversight: Data Monitoring Committee: No

SUMMARY:
Glioblastoma(GBM) is the most common malignant primary brain tumor and has unfortunately bad prognosis .PDL(Programmed death lignad 1)1 is alignad for a protein receptor PD1(Programmed death 1) that upon their engagement, an immunoinhibitory signal is generated thus allowing the tumor cells to evade the immune regulation and cytotoxic T lymphocytes(CTL). Also there have been many actions generated upon PDL1 binding with its receptor, among them is activation of autophagy that also serves for promoting tumor development and progression.Our study aims to detect PDL1 and LC3B levels in GBM , their relation with each other and the relation between their levels and overall survival of GBM cases.

DETAILED DESCRIPTION:
Gliomas account for almost 30% of all primary brain tumours, and are responsible for the majority of deaths from primary brain tumours .

Glioblastoma is the most common primary malignant brain tumor in adults, accounting for 60-70% of gliomas and 15% of primary brain tumors . Glioblastoma is the most aggressive and undifferentiated type of glioma and designated WHO Grade IV .

Programmed cell death 1 (PD-1) is a protein receptor that functions as an immune checkpoint. It conveys an inhibitory signal to T cells. In cancer, It protects tumors from cytotoxic T lymphocytes(CTL) . The inter¬action of PD1 with its ligand PD-L1 on surface of T-cells suppresses their function and hindering the recognition of tumor cells .PD-L1 expression is inversely correlated with the density of intratumoral CD8+(Cluster of Differentiation 8) T cells .

Autophagy is a catabolic process that leads to cellular degradation and recycling by lysosomal digestion. Thus allowing cells to adapt to stress). Autophagy promotes tumor development, progression and therapy resistance due to its pro-survival role under stress as radiation and chemotherapy. LC3B(microtubule associated protein light chain 3 B) is a commonly used marker to monitor autophagy .PD-L1 has been related to autophagy. Recent findings from experiments with murine melanoma cells and human ovarian cancer cells indicated cells expressing high levels of PD-L1 are more sensitive to autophagy inhibitors than cells that weakly express PD-L1. This finding provides potential opportunities for using autophagy inhibitors in PD-L1-overexpressing cells as a new avenue in cancer management . Thus not studied in GBM before ,our study is pure novel study.

The authors hypothesize that both PD-L1 and LC3B are highly expressed in GBM cells and high PDL1 expression is associated with low CTL count . It is possible that elevated levels of PD-L1 and LC3B markers indicate immune inhibition ,increased autophagy and poor prognosis thus their inhibition will have therapeutic benefit.

To date and to the best of our knowledge, this hypothesis has not been fully tested especially on our locality. To explore our hypothesis, this work is organized into three specific aims:

1. To evaluate relationship between PD-L1 expression and CTL count in GBM.
2. To evaluate the expression of PDL-1 and LC3B in GBM and to assess their relationship.
3. To explore the prognostic relevance of PDL-1 and LC3B in GBM by relating the level of their expression to some established prognostic factors (patient age, multifocal tumor, total or subtotal excision, tumor regrowth , karnofsky performance score and histopathological feature as: necrosis).

Formalin-fixed-paraffin-embedded tissue specimens of about sixty one cases of GBM and nearby apparently normal brain tissue will be obtained from private laboratory.

Histological diagnosis of H&E stained sections will be reviewed and the histological prognostic criteria will be assessed.

Immunohistochemical staining for PDL-1,CD8 and LC3B using mouse monoclonal antibodies with immunoperoxidase staining will be used as a visualization method. Antibodies dilutions, antigen retrieval methods, and incubation time will all be conducted according to the manufacturer's instructions.

Sample size calculation was carried out using G*Power 3 software . A calculated sample of 61 glioblastoma patients will be needed to detect an effect size of 0.1 (HR ranged between 1.54 and 1.74 in the multivariate Cox Hazard Proportion Regression for the PD-L1 expression level), with an error probability of 0.05 and 80% power on a one-tailed test.

Correlation between PD-L1 ,CTL count and LC3B expression and prognostic criteria of GBM will be performed using a computer software SPSS(Statistical Package for Social Sciences).

ELIGIBILITY:
Inclusion Criteria:

- Glioblastoma Multiforme patients with available follow up data

Exclusion Criteria:

* Specimens with no available follow up data

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: specimens of 61 cases will be obtained from the pathology laboratory of Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
This research will provide valuable insights into the pathogenesis of glioblastoma and the expression of PD-L1 &LC3B in this tumor especially in our locality. It will add to the literature a very important data regarding this field. | 2 years
  Evaluation of relationship between PD-L1,LC3B expression and CTL count in GBM. 2) Evaluation of the expression of PDL-1 and LC3B in GBM and assess their relationship.
  3) Exploration of the prognostic relevance of PDL-1 and LC3B in GBM by relating the level of their expression to some established prognostic factors (patient age, multifocal tumor, total or subtotal excision, tumor regrowth , and histopathological feature as: necrosis).

REFERENCES:
- [Background] Scobie MR, Houke HR, Rice CD. Modulation of glioma-inflammation crosstalk profiles in human glioblastoma cells by indirubin-3'-(2,3 dihydroxypropyl)-oximether (E804) and 7-bromoindirubin-3'-oxime (7BIO). Chem Biol Interact. 2019 Oct 1;312:108816. doi: 10.1016/j.cbi.2019.108816. Epub 2019 Sep 7. PMID 31505164
- [Background] Rahman M, Kresak J, Yang C, Huang J, Hiser W, Kubilis P, Mitchell D. Analysis of immunobiologic markers in primary and recurrent glioblastoma. J Neurooncol. 2018 Apr;137(2):249-257. doi: 10.1007/s11060-017-2732-1. Epub 2018 Jan 4. PMID 29302887